CLINICAL TRIAL: NCT01285817
Title: A Phase II Clinical Trial Using Metronomic Oral Low-dose Cyclophosphamide Alternating With Low-dose Oral Methotrexate With Continuous Celecoxib and Weekly Vinblastine in Children and Adolescents With Relapsed or Progressing Solid Tumours.
Brief Title: A Clinical Trial Using Metronomic Oral Low-dose Cyclophosphamide Alternating With Low-dose Oral Methotrexate With Continuous Celecoxib and Weekly Vinblastine in Children and Adolescents With Relapsed or Progressing soliD Tumours.
Acronym: SFCE METRO 01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12; 2010-021792-81 (EudraCT Number)
Record Dates: First submitted 2011-01-06; First posted 2011-01-28 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2015-10

CONDITIONS: Survival Without Progression
MeSH Terms: interventions — Celecoxib; Vinblastine; Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- traetment (Experimental)
  Interventions: Drug: celecoxib, Vinblastine, Cyclophosphamide , methotrexate ,

INTERVENTIONS:
Drug: celecoxib, Vinblastine, Cyclophosphamide , methotrexate ,

SUMMARY:
To establish the anti-tumour effect of this metronomic combination regimen defined by progression-free survival (PFS) after two cycles of treatment (4 months) and 12 months of treatment, as well as response rate after any number of cycles of treatment ("best response").

To define the safety profile of the combination. To characterize pharmacodynamics of the drug combination with the use of angiogenic markers (CEP, CEC, microparticles).

DETAILED DESCRIPTION:
Multi-center, combination phase II study, open-label, non-comparative, non-randomized.

All progressive or recurrent solid tumours will be included in the Phase II study, provided there are no curative options anymore.

Total expected number of patients (minimum maximum): 54 to 90 (2-stage design)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed malignant solid tumour.
* Progression or recurrence of the tumour radiologically established or confirmed within the 4 weeks prior to inclusion.
* Disease must be considered refractory to any line of conventional therapy or for which no effective conventional treatment exists.
* Age: ≥4 to 21 years of age at study entry
* Life expectancy: at least 8 weeks
* ECOG Performance status ≤ 1 or Lansky-Play Scale ≥ 70%
* Written informed consent of parent/guardian and patient assent
* Wash out of 4 weeks in case of prior chemotherapy, 6 weeks if treatment included nitrosoureas, 2 weeks in case of vincristine alone; 6 weeks in case of prior radiotherapy (except palliative radiotherapy on non measurable lesions).
* Patients must have recovered from the acute toxic effects of all prior therapy before enrolment into the study
* Able to comply with scheduled follow-up and with management of toxicity
* All patients with reproductive potential must practice an effective method of birth control while on study.
* Female patients aged > 12 years must have a negative pregnancy test within 7 days before study treatment.
* Capable of swallowing oral medication

Exclusion Criteria:

* Pregnant and breast feeding women.
* Uncontrolled intercurrent illness or active infection
* Inability to swallow oral medication.
* Patients on anticonvulsants will be allowed on study

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2011-01-12 (Actual); Primary Completion 2015-09-11 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Anti-tumour efficacy | 3 YEARS

SECONDARY OUTCOMES:
Safety AND Pharmacodynamic Study | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Verschuur A, Heng-Maillard MA, Dory-Lautrec P, Truillet R, Jouve E, Chastagner P, Leblond P, Aerts I, Honore S, Entz-Werle N, Sirvent N, Gentet JC, Corradini N, Andre N. Metronomic Four-Drug Regimen Has Anti-tumor Activity in Pediatric Low-Grade Glioma; The Results of a Phase II Clinical Trial. Front Pharmacol. 2018 Sep 27;9:00950. doi: 10.3389/fphar.2018.00950. eCollection 2018. PMID 30319400
- [Derived] Andre N, Abed S, Orbach D, Alla CA, Padovani L, Pasquier E, Gentet JC, Verschuur A. Pilot study of a pediatric metronomic 4-drug regimen. Oncotarget. 2011 Dec;2(12):960-5. doi: 10.18632/oncotarget.358. PMID 22156656